CLINICAL TRIAL: NCT02448641
Title: A Double-Blind, Controlled Phase 2b Study of the Safety and Efficacy of Modified Stem Cells (SB623) in Patients With Chronic Motor Deficit From Ischemic Stroke
Brief Title: Study of Modified Stem Cells (SB623) in Patients With Chronic Motor Deficit From Ischemic Stroke
Acronym: ACTIsSIMA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SanBio, Inc. (Industry)
Collaborators: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SB-STR02
Record Dates: First submitted 2015-05-15; First posted 2015-05-19 (Estimated); Results first posted 2020-04-17 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-04

CONDITIONS: Chronic Ischemic Stroke
Keywords: ischemic stroke; chronic stroke; fixed motor deficits
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- SB623 Implant (2.5M) (Experimental): 2.5 million SB623 cells
  Interventions: Biological: SB623 Implant (2.5M)
- SB623 Implant (5.0M) (Experimental): 5 million SB623 cells
  Interventions: Biological: SB623 Implant (5.0M)
- Sham Control (Sham Comparator): Sham surgery
  Interventions: Procedure: Sham surgery

INTERVENTIONS:
Biological: SB623 Implant (2.5M) — 2.5 million SB623 cells
  Arms: SB623 Implant (2.5M)
Biological: SB623 Implant (5.0M) — 5 million SB623 cells
  Arms: SB623 Implant (5.0M)
Procedure: Sham surgery
  Arms: Sham Control

SUMMARY:
Controlled study of stereotactic, intracranial injection of SB623 cells in patients with fixed motor deficits from ischemic stroke

DETAILED DESCRIPTION:
This is a double-blind, sham-surgery controlled study of stereotactic, intracranial injection of SB623 cells in patients with fixed motor deficits from ischemic stroke. The study will be conducted at approximately 65 sites in the United States.

Two cohorts, Group 1 (2.5 and 5 million SB623 cells combined) and Group 2 (sham placebo), will be included in this study. Subjects who are randomized into this study will receive either 2.5 million SB623 cells, 5 million SB623 cells or sham surgery at a 1:1:1 randomization ratio. Randomization will be performed via an interactive web/voice response system (IXRS), stratified by Screening mRS score (recorded in the IXRS at the clinical site).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years, inclusive
2. Documented history of completed ischemic stroke in subcortical region of MCA or lenticulostriate artery with or without cortical involvement, with correlated findings by MRI
3. Between 6 and 90 months (7.5 years) post-stroke, and having a chronic motor neurological deficit
4. Neurological motor deficit substantially due to incident stroke
5. Modified Rankin Score of 2-4
6. Require Motricity Index 30-75 (UE Scale) or 27-74 (LE Scale)
7. Able to undergo all planned neurological assessments
8. Able and willing to undergo magneti resonance imaging (MRI) with contrast and computed tomography (CT)
9. Agree that use of antiplatelet, anti-coagulant, or non-steroidal anti-inflammatory drugs to be determined by the local medical staff and in accordance with the ACCP 2012 guideline "Perioperative Management of Antithrombotic Therapy: Antithrombotic Therapy and Prevention of Thrombosis, 9th Edition: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines", if applicable , provided that no antiplatelet, anti-coagulant, or non-steroidal anti-inflammatory drugs are to be restarted post-surgery until after the Day 8 MRI is read and are determined to be safe to re-start
10. Subjects must have had physical therapy prior to entry (and be willing to continue to the extent possible)
11. Must be willing to discontinue herbal or non-traditional medicines for 1 week before and 1 week after the surgical procedure and be willing to continue to the extent possible
12. Ability of patient or legal authorized representative to understand and sign an Informed Consent

Exclusion Criteria:

1. History or presence of any other major neurological disease other than stroke
2. Cerebral infarct size >150 cm3 measured by MRI
3. Primary intracerebral hemorrhage
4. Myocardial infarction within prior 6 mos.
5. Malignancy unless in remission >5 yrs.
6. Clinically significant finding on MRI of brain not related to stroke
7. Any seizures in the 3 months prior to Screening
8. More than 5 degrees of contracture at shoulder, elbow, wrist, fingers, hip, knee and ankle
9. Other neurologic, neuromuscular or orthopedic disease that limits motor function
10. Uncontrolled systemic illness, including, but not limited to: hypertension; diabetes; renal, hepatic, or cardiac failure
11. Positive findings on tests for occult malignancy, unless a non-malignant etiology is confirmed
12. Uncontrolled major psychiatric illness, including depression symptoms (CESD R Scale of ≥16 is exclusionary)
13. Total bilirubin >1.9 mg/dL at Screening
14. Serum creatinine >1.5 mg/dL at Screening
15. Hemoglobin <10.0 g/dL at Screening
16. Absolute neutrophil count <2000 /mm3 at Screening
17. Absolute lymphocytes <800 /mm3 at Screening
18. Platelet count <100,000 /mm3 at Screening
19. Liver disease supported by AST (SGOT) or ALT (SGPT) ≥2.5 x upper limit of normal at Screening
20. Serum calcium >11.5 mg/dL at Screening
21. International Normalized Ratio of Prothrombin Time (INR) >1.2 at Screening if the patient does not take anticoagulants; for patients on anticoagulants, INR must be confirmed to be ≤1.2 prior to surgery
22. Presence of craniectomy or other contraindication to stereotactic surgery
23. Participation in any other investigational trial within 4 weeks of initial screening and within 7 weeks of Baseline visit
24. Botulinum toxin injection, phenol injection, intrathecal baclofen, or any other interventional treatments for spasticity (except bracing and splinting) 16 weeks prior to the Baseline visit
25. Substance use disorder (per DSM-V criteria, including drug or alcohol)
26. Contraindications to head MRI (with constrast) or CT
27. Pregnant or lactating
28. Female patients of childbearing potential unwilling to use an adequate birth control method during the 12 months of the study
29. Any other condition or situation that the investigator believes may interfere with the safety of the subject or the intent and conduct of the study
30. Any prior SB623 cell implantation and/or any prior stem cell treatment for stroke or other reason regardless of mode of administration

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2016-03-08 (Actual); Primary Completion 2018-12-05 (Actual); Study Completion 2018-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Steinberg, MD, PhD, Principal Investigator — Stanford Hospital and Clinics, School of Medicine
Locations (65):
- United States (65):
  - University of Alabama at Birmingham (Surgical/Assessment), Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Xenoscience, Inc. (Assessment), Phoenix, Arizona
  - The Research Center of Southern California (Assessment), Carlsbad, California
  - Rancho Los Amigos National Rehab Center, Downey, California
  - Neuro-Pain Medical Center (Assessment), Fresno, California
  - Neuro Pain Medical Center, Fresno, California
  - University of California Irvine, Irvine, California
  - Ronald Reagan UCLA Medical Center (Assessment/Surgical), Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - University of California Irvine (Assessment), Orange, California
  - Westview Clinical Research (Assessment), Placentia, California
  - Providence Saint John's Health Center (Assessment), Santa Monica, California
  - Providence St. John's Health Center (Surgical), Santa Monica, California
  - Providence St. Johns Health Center, Santa Monica, California
  - Stanford Health Care (Surgical/Assessment), Stanford, California
  - New England Institute for Clinical Research (Assessment), Stamford, Connecticut
  - MedStar National Rehabilitation Hospital (Assessment), Washington D.C., District of Columbia
  - University of Miami Miller School of Medicine (Assessment/Surgical), Miami, Florida
  - University of Miami Jackson Memorial Hospital, Miami, Florida
  - NeuroMedical Research Institute (Assessment), Panama City, Florida
  - Medsol Clinical Research Center (Assessment), Port Charlotte, Florida
  - Neurostudies, Inc. (Assessment), Port Charlotte, Florida
  - University of South Florida (Assessment), Tampa, Florida
  - Grady Memorial Hospital (Assessment), Atlanta, Georgia
  - Emory University Hospital (Surgical), Atlanta, Georgia
  - Center for Advanced Research and Education (Assessment), Gainesville, Georgia
  - Northwestern Memorial Hospital (Surgical), Chicago, Illinois
  - University of Chicago Medical Center (Assessment), Chicago, Illinois
  - University of Chicago Medical Center (Surgical), Chicago, Illinois
  - Rehabilitation Institute of Chicago, Chicago, Illinois
  - Consultants in Neurology, Ltd. (Assessment), Northbrook, Illinois
  - OSF Saint Francis Healthcare System (Assessment), Peoria, Illinois
  - Indiana Medical Research, Elkhart Clinic (Assessment), Elkhart, Indiana
  - University of Kansas Medical Center (Surgical), Kansas City, Kansas
  - Kansas Institute of Research (Assessment), Overland Park, Kansas
  - University of Kentucky Hospital (Surgical), Lexington, Kentucky
  - University of Louisville Clinical Trials Unit (Assessment), Louisville, Kentucky
  - NeuroMedical Clinic of Central Louisiana (Assessment), Alexandria, Louisiana
  - Beth Israel Deaconess Medical Center (Surgical), Boston, Massachusetts
  - Wayne State University (Assessment), Detroit, Michigan
  - Henry Ford Health System (Assessment), Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Rutgers New Jersey Medical School (Assessment), Newark, New Jersey
  - New York University Langone Medical Center (Surgical/Assessment), New York, New York
  - NYU Langone Medical Center, New York, New York
  - The Burke Rehabilitation Hospital (Assessment), White Plains, New York
  - Carolinas Rehabilitation (Assessment), Charlotte, North Carolina
  - Neurology and Neuroscience Associates, Inc. (Assessment), Akron, Ohio
  - Neurology and Neuroscience Associates, Akron, Ohio
  - University Hospital Case Medical Center (Surgical), Cleveland, Ohio
  - University of Toledo Medical Center (Assessment), Toledo, Ohio
  - Moss Rehab (Assessment), Elkins Park, Pennsylvania
  - Hospital of the University of Pennsylvania (Assessment), Philadelphia, Pennsylvania
  - Pennsylvania Hospital (Surgical), Philadelphia, Pennsylvania
  - Thomas Jefferson University Comprehensive Stroke Center (Assessment), Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center (Surgical/Assessment)), Pittsburgh, Pennsylvania
  - Abington Neurological Associates (Assessment), Willow Grove, Pennsylvania
  - Medical University of South Carolina (Surgical), Charleston, South Carolina
  - Chattanooga Center for Neurologic Research (Assessment), Chattanooga, Tennessee
  - University of Texas Medical School, Dallas, Texas
  - University of Texas Health Science Center at Houston (Assessment/Surgical), Houston, Texas
  - West Virginia University Hospitals (Assessment), Morgantown, West Virginia
  - West Virginia University, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Sham Control: Control Group: Sham surgery
Period: Overall Study
Arm/Group | SB623 Implant (2.5M) | SB623 Implant (5.0M) | Sham Control
Started | 55 | 56 | 52
Completed | 54 | 51 | 48
Not Completed | 1 | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SB623 Implant (2.5M) | SB623 Implant (5.0M) | Sham Control | Total
Number analyzed (Participants) | 55 | 56 | 52 | 163
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.5 (11.08) | 58.9 (9.99) | 55.2 (11.57) | 57.2 (10.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 20 | 19 | 60
  Male | 34 | 36 | 33 | 103
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 0 | 6
  Not Hispanic or Latino | 52 | 53 | 52 | 157
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 1 | 2 | 6 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 6 | 1 | 2 | 9
  White | 45 | 51 | 42 | 138
  Other | 3 | 2 | 1 | 6
Region of Enrollment [Number; unit: participants]
  United States | 55 | 56 | 52 | 163

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Whose Fugl-Meyer Motor Total Score (FMMS) Improved by ≥ 10 Points at Month 6 From Baseline
Description: The FMMS is used as a clinical measure of body function impairment after stroke that assesses several dimensions of motor impairment, including range of motion in both upper and lower limbs, reflex activity, volitional movement, and co-ordination.
  The FMMS motor component consists of the 33-item upper extremity subscale (UE-FMMS) and the 17-item lower extremity subscale (LE-FMMS). Items were scored on a 3-point ordinal scale:
  0= cannot perform; 1= partial motion; 2= full motion
  Individual items were then summed to determine scores for the 2 subscale scores, as well as a motor total score (total of all item scores including the 2 subscales UE-FMMS and LE-FMMS). As a result, the UE-FMMS subscale score ranged from 0 to 66 and the LE-FMMS subscale score ranged from 0 to 34. The FMMS motor total score ranged from 0 (hemiplegia) to a maximum of 100 points (normal motor performance).
  Responders: subjects whose FMMS motor total score improve by ≥10 points at Month 6 from Baseline
Time Frame: 6 months
Population: Modified Intent-to-Treat (mITT) Population: Included all randomized subjects who completed the surgery treatment procedure. A total of 111 subjects received treatment with SB623; 55 subjects were randomized to receive 2.5 million SB623 cells and 56 subjects to receive 5 million SB623 cells.
Measure: Count of Participants; unit: Participants
Arm/Group | SB623 Implant (2.5M) | SB623 Implant (5.0M) | Sham Control
Number analyzed (Participants) | 55 | 56 | 52
Participants
  Responder | 7 | 9 | 7
  Non-responder | 46 | 45 | 38
  Unknown | 2 | 2 | 7
Statistical Analysis 1: Comparison: SB623 Implant (2.5M) vs SB623 Implant (5.0M) vs Sham Control; Combined SB623 Implant Vs Sham Surgery group at Month 6; Test type: Superiority; p = 0.6743, Mixed Models Analysis — GLMM: Generalized Linear Mixed Model; A GLMM with FMMS responder as outcome, treatment, visit, treatment-visit interaction, pooled site, Baseline FMMS and Baseline mRS scores as covariates; Odds Ratio (OR) = 1.33, 95% CI 2-sided [0.35 to 5.09]

2. Secondary Outcome: Modified Rankin Scale Response: The Proportion of Subjects That Improved at Least One Point on the mRS From Baseline
Description: Responders: The subjects that improved at least one point on the mRS from Baseline
  Modified Rankin Scale (mRS): This scale is used to measure the degree of disability or dependence in the daily activities of people who had suffered a stroke. The mRS is an ordinal scale from 0 (no symptoms at all) to 5 (severe disability; requiring constant nursing care and attention, bedridden, incontinent) with a sixth category of death.
Time Frame: 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Sham Control: Sham surgery Group
Arm/Group | SB623 Implant (2.5M) | SB623 Implant (5.0M) | Sham Control
Number analyzed (Participants) | 55 | 56 | 52
Participants
  Responder | 6 | 10 | 9
  Non-responder | 43 | 42 | 35
  Unknown | 6 | 4 | 8
Statistical Analysis 1: Comparison: SB623 Implant (2.5M) vs SB623 Implant (5.0M) vs Sham Control; Combined SB623 Implant Vs Sham Surgery group at Month 6; Test type: Superiority; p = 0.1000, Mixed Models Analysis — GLMM: Generalized Linear Mixed Model; A GLMM with mRS responder as outcome, treatment, visit, treatment-visit interaction, pooled site and Baseline mRS scores as covariates; Odds Ratio (OR) = 0.43, 95% CI 2-sided [0.15 to 1.18]

3. Secondary Outcome: The Proportion of Subjects That Improved at Least 6 Points From Baseline on the ARAT Total Score at the Affected Side
Description: Responders: The subjects that improved at least 6 points from Baseline on the ARAT total score at the affected side.
  Action Research Arm Test (ARAT): The test was scored for left and right side separately. Performance on each item was rated on a 4-point ordinal scale ranging from: 3 (performed test normally in less than 5 seconds); 2 (completed test, but took abnormally long or had great difficult, with time varying from 5 to 60 seconds; 1 (performed test partially); 0 (could perform no part of the test). The ARAT is a 19-item measure divided into 4 subtests: Grasp subscale (with 6 items and a score range of 0 to 18); Grip subscale with 4 items and a score range of 0 to 12); Pinch subscale with 6 items and a score range of 0 to 18); Gross arm movement subscale (with 3 items and a score range of 0 to 9). The maximum score on the ARAT is 57 points (possible range 0 to 57) for each side.
Time Frame: 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Sham Control: Sham surgery Group (Control)
Arm/Group | SB623 Implant (2.5M) | SB623 Implant (5.0M) | Sham Control
Number analyzed (Participants) | 55 | 56 | 52
Participants
  Responder | 6 | 9 | 9
  Non-responder | 47 | 45 | 37
  Unknown | 2 | 2 | 6

4. Secondary Outcome: The Proportion of Subjects That Improved at Least 1 Functional Level From Baseline on Gait Velocity
Description: Responders: The subjects that improved at least 1 functional level (eg, from < 0.4 m/s to 0.4-0.8 m/s or from 0.4-0.8 m/s to > 0.8 m/s) from Baseline on Gait Velocity.
  Gait Velocity was measured on a standard 10 meter walk. Two trials were tested and the average result from both was used for analysis
Time Frame: 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SB623 Implant (2.5M) | SB623 Implant (5.0M) | Sham Control
Number analyzed (Participants) | 55 | 56 | 52
Participants
  Responder | 7 | 6 | 5
  Non-respinder | 39 | 43 | 36
  Unknown | 9 | 7 | 11

5. Secondary Outcome: Neurological Quality of Life Response: T-scores of the Change From Baseline in the 2 Sub-domains (Upper Extremity Function and Lower Extremity Function)
Description: The Neurological Quality of Life (NeuroQOL) was used as a measure of change in the levels of Quality of Life, Satisfaction and Participation, secondary to improvements in the subject's upper and lower extremity motor function. NeuroQOL is summation of item scores for upper extremity (8 terms: score 8 - 40) and lower extremity (8 items: score 8 - 40) separately. The item scores are on a 1 to 5 scale (1 = unable to do; 2 = with much difficulty; 3 = with some difficulty; 4 = with little difficulty; 5 = without any difficulty). The result provided here shows NeuroQOL score converted to T-score. The range for Upper extremity T-score and Lower extremity T-score are 12.8 to 53.8 and 16.5 to 58.6 respectively.
Time Frame: 6 Months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Change in score on a scale from baseline
Groups:
- SB623 Implant (2.5 M): 2.5 million SB623 cells SB623 Implant (2.5M): 2.5 million SB623 cells
- SB623 Implant (5.0M): 5.0 million SB623 cells SB623 Implant (5.0M): 5.0 million SB623 cells
- Sham Surgery: Sham surgery: Control Group
Arm/Group | SB623 Implant (2.5 M) | SB623 Implant (5.0M) | Sham Surgery
Number analyzed (Participants) | 55 | 56 | 52
Change in score on a scale from baseline
  Upper Extremity Function | 0.14 (2.018) | -1.08 (2.000) | -0.11 (1.946)
  Lower Extremity Function | 1.61 (1.343) | 2.74 (1.331) | 1.60 (1.301)
Statistical Analysis 1: Comparison: SB623 Implant (2.5 M) vs SB623 Implant (5.0M) vs Sham Surgery; Statistical analysis: NeuroQOL score for the Upper Extremity Function (Represents Mean Change from Baseline in T-Scores at Month 6); Test type: Superiority; p = 0.7788, Mixed Models Analysis — Combined SB623 vs. Sham at month 6 MMRM: Mixed Model for Repeated Measures; MMRM included treatment, visit, pooled site, corresponding Baseline sub-domain T-score, Baseline mRS score, and the treatment-by-visit interaction; Mean Difference (Net) = -0.36, 95% CI 2-sided [-2.90 to 2.17] — LSMD (Least square mean difference) (SE): -0.36 (1.283)
Statistical Analysis 2: Comparison: SB623 Implant (2.5 M) vs SB623 Implant (5.0M) vs Sham Surgery; Statistical Analysis: NeuroQOL score for Lower Extremity Function (Represents Mean Change from Baseline in T-Scores at Month 6); Test type: Superiority; p = 0.5347, Mixed Models Analysis — Combined SB623 vs. Sham at month 6 MMRM: Mixed Model for Repeated Measures; [statistical method as in outcome 5, analysis 1]; Mean Difference (Net) = 0.58, 95% CI 2-sided [-1.26 to 2.43] — LSMD (Least square mean difference) (SE): 0.58 (0.934)

6. Secondary Outcome: Global Rating of Perceived Change (GRPC): The Proportion of Subjects Scoring Either 7 or 6 on the Global Rating of Perceived Change by Both Subject and Clinician
Description: Responders: Participants who scored either 7 [much better] or 6 [a little better, meaningful])
  Global Rating of Perceived Change from Baseline: Subjects and Clinicians were asked about perceived changes in their motor function by comparing "how well they are doing compared to before the surgical procedure". The Subject Global Rating of Perceived Change was completed by the subject (or by the caregiver using the subject's answers). The following 7-point Likert scale was used: Score 7 (much better); Score 6 (a little better, meaningful); Score 5 (a little better, not meaningful); Score 4 (about the same); Score 3 (a little worse, not meaningful); Score 2 (a little worse, meaningful); Score 1 (much worse)
Time Frame: 6 Months (LOCF)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SB623 Implant (2.5M) | SB623 Implant (5.0M) | Sham Control
Number analyzed (Participants) | 55 | 56 | 52
Participants
  As per Clinician: Responder | 15 | 18 | 13
  As per Clinician: Non-responder | 39 | 38 | 39
  As per Clinician: Unknown | 1 | 0 | 0
  As per Subject: Responder | 18 | 25 | 22
  As per Subject: Non-responder | 37 | 31 | 30
  As per Subject: Unknown | 0 | 0 | 0

7. Other Pre Specified Outcome: Additional Analysis (MMRM), Fugl-Meyer Motor Scale (FMMS)
Description: An additional analysis using mixed model for repeated measures (MMRM) was performed treating the change from Baseline in FMMS total score as a continuous outcome (dependent) variable. The independent variables were treatment, visit, treatment-by-visit interaction, and pooled surgical site as effects, and Baseline FMMS total score and Baseline mRS score as covariates. Least-squares means (LS-mean) with SE was calculated for the change from baseline measurements.
Time Frame: 6 Months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Change in score on a scale from baseline
Arm/Group | SB623 Implant (2.5 M) | SB623 Implant (5.0M) | Sham Surgery
Number analyzed (Participants) | 55 | 56 | 52
Change in score on a scale from baseline | 5.3 (1.64) | 4.5 (1.62) | 3.6 (1.59)
Statistical Analysis 1: Comparison: SB623 Implant (2.5 M) vs SB623 Implant (5.0M) vs Sham Surgery; Change from Baseline at Month 6 Between-group Effect size is calculated as the LS mean difference divided by the model estimate of the pooled SD, obtained from the square root of the diagonal element, associated with the analysis visit summarized, from the covariance matrix; Test type: Superiority; p = 0.2959, Mixed Models Analysis — MMRM: Mixed effect Model Repeat Measurement; [statistical method as in outcome 5, analysis 1]; Mean Difference (Net) = 1.2, 95% CI 2-sided [-1.1 to 3.6] — LSMD (Least square mean difference) (SE): 1.2 (1.18)

8. Other Pre Specified Outcome: Proportion of Subjects Whose FMMS Motor Total Score Improve by ≥10 Points at Month 6 From Baseline (Per Protocol Population)
Description: Responders: subjects whose FMMS motor total score improve by ≥10 points at Month 6 from Baseline
Time Frame: Month 6
Population: Per Protocol (PP) Population: The PP population included all subjects in the mITT population who did not have important protocol deviations.
Measure: Count of Participants; unit: Participants
Arm/Group | SB623 Implant (2.5M) | SB623 Implant (5.0M) | Sham Control
Number analyzed (Participants) | 41 | 46 | 46
Participants
  Responder | 6 | 9 | 7
  Non-responder | 34 | 35 | 35
  Unknown | 1 | 2 | 4
Statistical Analysis 1: Comparison: SB623 Implant (2.5M) vs SB623 Implant (5.0M) vs Sham Control; Combined SB623 Implant Vs Sham Surgery group at Month 6; Test type: Superiority; p = 0.6854, Mixed Models Analysis — GLMM: Generalized Linear Mixed Model; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.36, 95% CI 2-sided [0.31 to 5.92]

ADVERSE EVENTS:
Time Frame: Safety was monitored throughout the study. The adverse event reporting period for this trial began upon informed consent and ended 12 months after the administration of SB623, or at Early Termination. Also, an external Data Safety Monitoring Board (DSMB) was utilized to review safety data, including clinical symptoms, laboratory findings, and MRI brain imaging. The DSMB reviewed study data within one month of the enrollment of subjects at the 25%, 50%, and 75% of the total population.
Groups:
- Sham Control: Control Group: Sham surgery Group
Arm/Group | SB623 Implant (2.5M) | SB623 Implant (5.0M) | Sham Control
All-Cause Mortality (participants affected / at risk) | 0/55 | 1/56 | 0/52
Serious Adverse Events (participants affected / at risk) | 15/55 | 15/56 | 10/52
Other Adverse Events (participants affected / at risk) | 52/55 | 53/56 | 51/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SB623 Implant (2.5M) (N=55) | SB623 Implant (5.0M) (N=56) | Sham Control (N=52)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (3) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (2) | 0 (0) | 1 (1)
Pancreas infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchopneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Intervertebral discitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Crush injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Incision site complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Pneumocephalus (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Anti factor X antibody positive (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 4 (4) | 4 (5) | 3 (4)
Basal ganglia haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure like phenomena (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SB623 Implant (2.5M) (N=55) | SB623 Implant (5.0M) (N=56) | Sham Control (N=52)
Eye swelling (Eye disorders) | 3 (3) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 13 (13) | 12 (12) | 3 (3)
Vomiting (Gastrointestinal disorders) | 10 (10) | 6 (6) | 1 (1)
Constipation (Gastrointestinal disorders) | 5 (5) | 2 (2) | 4 (5)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1)
Fatigue (General disorders) | 3 (3) | 3 (3) | 4 (4)
Pyrexia (General disorders) | 1 (1) | 3 (3) | 1 (1)
Pain (General disorders) | 0 (0) | 3 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (3) | 5 (5) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 4 (5) | 2 (2)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2) | 3 (3)
Procedural headache (Injury, poisoning and procedural complications) | 8 (9) | 9 (9) | 13 (13)
Procedural pain (Injury, poisoning and procedural complications) | 11 (11) | 5 (5) | 6 (6)
Fall (Injury, poisoning and procedural complications) | 5 (8) | 5 (5) | 4 (12)
Incision site pain (Injury, poisoning and procedural complications) | 5 (5) | 5 (5) | 10 (10)
Contusion (Injury, poisoning and procedural complications) | 2 (4) | 3 (3) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) | 5 (5)
Headache (Nervous system disorders) | 35 (42) | 41 (48) | 32 (35)
Paraesthesia (Nervous system disorders) | 1 (1) | 3 (4) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 3 (5) | 1 (1)
Depression (Psychiatric disorders) | 6 (7) | 3 (3) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 2 (3) | 2 (2) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-01-05): https://cdn.clinicaltrials.gov/large-docs/41/NCT02448641/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-21): https://cdn.clinicaltrials.gov/large-docs/41/NCT02448641/SAP_001.pdf